CLINICAL TRIAL: NCT06435091
Title: REBECCA-3 Study, Research on Breast Cancer Induced Chronic Conditions Supported by Causal Analysis of Multi-source Data
Acronym: REBECCA-3
Status: Active, not recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: REBECCA3SUH; REBECCA-PROST (Other: European Union's Horizon 2020); 965231 (Other Grant/Funding Number: European Union's Horizon 2020)
Record Dates: First submitted 2024-03-14; First posted 2024-05-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cancer Related Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overall aim of the REBECCA project is to exploit the potential of "real-world data" to support clinical research and improve existing clinical workflow. The primary aim of the REBECCA-3 study is to use multi-source "real-world data" to monitor the quality of life (QoL) of prostate cancer patients who are affected by cancer-related fatigue during and after treatment. This is to investigate whether the REBECCA monitoring is accepted by male patients and can be used within various forms of cancer.

Study design: 40 prostate cancer patients that undergo radiology and/or chemotherapy treatment will be included at the time of diagnosis. After end of primary treatment, the patients will receive a smartwatch, and have to download a REBECCA patient app on their mobile and a PC plug-in on their PC so that we can monitor their QoL for 4 months. In addition to collecting digital QoL parameters through the REBECCA-system, patient-reported QoL measures will also be collected through standardized PROMs and self-evaluation forms. Further, biological samples (blood, urine, and faeces) are collected at three time points of the study (i.e., at the time of: diagnosis, completed treatment, and 4 months post treatment), to investigate immunologic biomarkers, DNA methylation patterns and microbiota for assessment of new biological and prognostic information related to the development of cancer-related fatigue in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients with histologically detectable M0 prostate cancer requiring primary surgery or primary radiation therapy followed by hormone therapy at least and no more than 3 months of initiation prior to study start
* Male prostate cancer patients under 80 years of age.
* Patients who have an increased life expectancy beyond the first 3 months after starting treatment.
* Patients who have the ability to understand the protocol and can participate in the follow-up plan.
* Patients who have the absence of psychological, familial, sociological, or geographic condition potentially hindering compliance with the study protocol and follow-up schedule.
* Patients who have a smart phone.

Exclusion Criteria:

* Patients who do not consent to the study protocol.
* Patients with a previous cancer diagnosis (except skin cancer treated only by surgery).
* Patients who have previously been treated with any form of chemotherapy/radiotherapy.
* Foreign-language patients without sufficient Norwegian understanding
* Patients who do not have a smartphone

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Prostate cancer patients at Stavanger University Hospital, Norway
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the average REBECCA system usage rate throughout the monitoring period. | From the end of treatment to the 4-month post-treatment follow-up.
  Daily and weekly frequency of participant interactions with the REBECCA system.

SECONDARY OUTCOMES:
Quality of life (QoL) measured by the EORTC-QLQ-C30. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ) C30 scores patients QoL on a scale of 0-100, where higher values indicate higher QoL.
Quality of life (QoL) measured by the SF36-questionnaire. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The SF36 scores the patients physical and mental health on a scale of 0-100, where higher values indicate better health.
Quality of life (QoL) measured by the EPIC-26-questionnaire. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The Expanded Prostate Cancer Index Composite short form 26 (EPIC-26) scores the patients QoL on a scale of 0-100, where higher values indicate better health.
Fatigue in primary prostate cancer patients measured by the fVAS questionnaire. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The fatigue Visual Analog Scale (fVAS) scores fatigue on a scale of 0-100, where lower values indicate less fatigue, thus a reduction in fVAS score between timepoints indicates a reduction of fatigue.
Fatigue in primary prostate cancer patients measured by the FSS questionnaire. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The Fatigue Severity Scale (FSS) scores fatigue on a scale of 1-7, where lower values indicate less fatigue, thus a reduction in FSS score between timepoints indicates a reduction of fatigue.
Fatigue in primary prostate cancer patients measured by the FQ questionnaire. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  The Fatigue Questionnaire (FQ) scores fatigue on a scale of 0-33, where lower values indicate less fatigue, thus a reduction in FQ score between timepoints indicates a reduction of fatigue.
REBECCA system index score | At the 4-month post-treatment follow-up.
  The REBECCA system index score is given as values between 0 and 100, where higher values indicate higher QoL.
Longitudinal analysis of the effect of the use of REBECCA using Generalized Estimating Equation (GEE) | From the end of treatment to the 4-month post-treatment follow-up.
  Weekly measurements over a 4-month period.
Fatigue biomarkers in plasma of primary prostate cancer patients. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  Measure levels of fatigue biomarkers: HSP90, IL1β, IL6, IL10, IL1βRa, and DNA methylation.
Gut microbiota composition in primary prostate cancer patients. | At the time of inclusion, at the end of treatment (3-6 months from time of inclusion) and at the 4-month post-treatment follow-up
  Long-read 16S rRNA sequencing of faecal samples to characterize the gut microbiota composition.
Correlation between the REBECCA system index score and QoL questionnaire scores. | At the 4-month post-treatment follow-up.
  REBECCA score (scale 0-100) correlation to the EORTC-QLQ-C30 (scale 0-100), SF36 (scale 0-100), and EPIC-26 (scale 0-100).
Correlation between the REBECCA system index score and fatigue questionnaire scores. | At the 4-month post-treatment follow-up.
  REBECCA score (scale 0-100) correlation to the fVAS (scale 0-100), FSS (scale 0-7) and FQ (scale 0-33).
Correlation between the REBECCA system index score and fatigue biomarker levels in plasma | At the 4-month post-treatment follow-up.
  REBECCA score (scale 0-100) correlation to fatigue biomarker levels of HSP90, IL1β, IL6, IL10, IL1βRa and DNA methylation in plasma.
Correlation between the REBECCA system index score and fatigue biomarker levels in feces. | At the 4-month post-treatment follow-up.
  REBECCA score (scale 0-100) correlation to fatigue biomarker levels of pro-inflammatory and anti-inflammatory microbes in feces.
Subjective assessments of system usability measured by the System Usability Scale questionnaire. | At the 4-month post-treatment follow-up.
  The System Usability Scale measures user satisfaction on a scale from 0-100, where a score >75 indicate system use satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, PhD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Stensland M, Bru KF, Austdal M, Dahl IH, Jonsdottir K, Lende TH, Heimvik C, Elve I, Omdal R, van der Giezen M, Kvivik I, Tangeland B, Davidsen L, Hashemi M, Cais A, van Dijk KJ, Seyoum Y, Blafjelldal V, Sola ST, Papadopoulos A, Kiriakidou N, Ioakeimidis I, Diou C, Sarafis I, Delopoulos A, Janssen EAM, Gilje B, Tjensvoll K. Monitoring cancer-related fatigue and quality of life in breast and prostate cancer patients after primary treatment: a study protocol for the REBECCA trials in Norway. Clin Exp Med. 2026 Feb 8;26(1):133. doi: 10.1007/s10238-026-02073-y. PMID 41655181
- See also: REBECCA Project Site — https://rebeccaproject.eu/